CLINICAL TRIAL: NCT01084356
Title: Evaluation of a New CZT System for Imaging in Routine Nuclear Medicine Examination
Brief Title: Evaluation of a New CZT System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Einat Even-Sapir MD, PhD. Head, Dept of Nuclear Medicine, Tel Aviv SoUrasky medical center
Other Study IDs: TASMC-10-EES-0649-CTIL
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Parathyroid Adenoma; Thyroid Adenoma
Keywords: CZT; sentinel node; osseous processes
MeSH Terms: conditions — Parathyroid Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- hand: patients admitted for Tc MDP for evaluation of carpal/metacarpal and finger bone lesions
- thyroid: patients admitted for Tc thyroid scan
- parathyroid: patients investigated for parathyroid adenoma
- sentinel node: patients who are due to sentinel node biopsy

SUMMARY:
The purpose of the study is to check if the new CZT system has an advantage in detection of small osseous processes, thyroid adenomas, parathyroid adenomas and detection of sentinel node, in comparison with the techniques in use.

Participants: 100 subjects male and female that come to the institute of nuclear medicine for routine screening examinations.

The CZT screening takes 10 minutes and does not require any extra intervention to the routine screening.

ELIGIBILITY:
Inclusion Criteria:

* age over 18

Exclusion Criteria:

* pregnancy
* patients unable to understand and sign an informed consent
* age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consequtive patiants admitted for the above scans and consented to be further investigated by the CZT system
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even Sapir, PhD, MD, Principal Investigator — Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Gambhir SS, Berman DS, Ziffer J, Nagler M, Sandler M, Patton J, Hutton B, Sharir T, Haim SB, Haim SB. A novel high-sensitivity rapid-acquisition single-photon cardiac imaging camera. J Nucl Med. 2009 Apr;50(4):635-43. doi: 10.2967/jnumed.108.060020. PMID 19339672
- [Background] Hruska CB, Phillips SW, Whaley DH, Rhodes DJ, O'Connor MK. Molecular breast imaging: use of a dual-head dedicated gamma camera to detect small breast tumors. AJR Am J Roentgenol. 2008 Dec;191(6):1805-15. doi: 10.2214/AJR.07.3693. PMID 19020253
- [Background] Mueller B, O'Connor MK, Blevis I, Rhodes DJ, Smith R, Collins DA, Phillips SW. Evaluation of a small cadmium zinc telluride detector for scintimammography. J Nucl Med. 2003 Apr;44(4):602-9. PMID 12679406
- [Background] Ketchum LE. New equipment in nuclear medicine, part 1: solid-state detectors. J Nucl Med. 1998 Nov;39(11):15N, 35N-36N. No abstract available. PMID 9829562
- [Background] Rhodes DJ, O'Connor MK, Phillips SW, Smith RL, Collins DA. Molecular breast imaging: a new technique using technetium Tc 99m scintimammography to detect small tumors of the breast. Mayo Clin Proc. 2005 Jan;80(1):24-30. doi: 10.1016/S0025-6196(11)62953-4. PMID 15667025
- [Background] O'Connor MK, Phillips SW, Hruska CB, Rhodes DJ, Collins DA. Molecular breast imaging: advantages and limitations of a scintimammographic technique in patients with small breast tumors. Breast J. 2007 Jan-Feb;13(1):3-11. doi: 10.1111/j.1524-4741.2006.00356.x. PMID 17214787
- [Background] Tsuchimochi M, Hayama K, Oda T, Togashi M, Sakahara H. Evaluation of the efficacy of a small CdTe gamma-camera for sentinel lymph node biopsy. J Nucl Med. 2008 Jun;49(6):956-62. doi: 10.2967/jnumed.108.050740. Epub 2008 May 15. PMID 18483107